CLINICAL TRIAL: NCT01477346
Title: Arthritis Research UK Gout Treatment Trial. Phase 2: Two Year Randomised Controlled Trial of a Nurse Led Package of Care
Brief Title: Arthritis Research UK Gout Treatment Trial - Phase 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Arthritis Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11115
Record Dates: First submitted 2011-11-14; First posted 2011-11-22 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse intervention (Other): Nurse led package of care based on current recommended best practice.
  Interventions: Other: Nurse intervention
- Standard care (Other): Continuing standard general practitioner led care
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Nurse intervention — Complex package of care involving patient information and advice concerning lifestyle modification and recommended drug therapy.
  Arms: Nurse intervention
Other: Standard care — Continuing standard General Practitioner led care.
  Arms: Standard care

SUMMARY:
The purpose of this study is to determine in community-derived patients with gout the effectiveness, and cost effectiveness, of a nurse-led complex intervention that reflects recommended best practice (including patient information concerning gout, its prognosis and its non-pharmacological and drug options).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gout
* At least one acute attack of gout within previous 12 months

Exclusion Criteria:

- Inability to give informed consent and known terminal or mental illness

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2013-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Reduction in serum uric acid levels | 2 years

SECONDARY OUTCOMES:
Reduction in number of self reported acute attacks during year 2 | 2 years
Improved Quality of Life scores at study end | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Doherty, MA MD FRCP, Principal Investigator — University of Nottingham
Locations (1):
- Academic Rheumatology, University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stamp LK, Frampton C, Morillon MB, Taylor WJ, Dalbeth N, Singh JA, Doherty M, Zhang W, Richardson H, Sarmanova A, Christensen R. Association between serum urate and flares in people with gout and evidence for surrogate status: a secondary analysis of two randomised controlled trials. Lancet Rheumatol. 2022 Jan;4(1):e53-e60. doi: 10.1016/S2665-9913(21)00319-2. Epub 2021 Nov 5. PMID 38288731
- [Derived] Doherty M, Jenkins W, Richardson H, Sarmanova A, Abhishek A, Ashton D, Barclay C, Doherty S, Duley L, Hatton R, Rees F, Stevenson M, Zhang W. Efficacy and cost-effectiveness of nurse-led care involving education and engagement of patients and a treat-to-target urate-lowering strategy versus usual care for gout: a randomised controlled trial. Lancet. 2018 Oct 20;392(10156):1403-1412. doi: 10.1016/S0140-6736(18)32158-5. PMID 30343856